CLINICAL TRIAL: NCT05050474
Title: A Clinical Study to Evaluate the Immunogenicity and Safety of the Third Dose Booster Immunization of Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01) in Healthy Participants
Brief Title: Booster Immunization Study of Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Collaborators: Guangdong Center for Disease Prevention and Control (Other Government); Simoon Record Pharma Information Consulting Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V-01-I-Booster
Record Dates: First submitted 2021-09-13; First posted 2021-09-20 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- V-01 COVID-19 Vaccine (Experimental): One dose administrated by intramuscular injection
  Interventions: Biological: Recombinant SARS-CoV-2 Fusion Protein Vaccine

INTERVENTIONS:
Biological: Recombinant SARS-CoV-2 Fusion Protein Vaccine — The product should be a milky-white suspension for injection. For prevention of SARS-CoV-2 infection.
  Other Names: V-01

SUMMARY:
This study is a continuation study of the original V-01-I phase trial, using a single-center, single-arm, open design to evaluate the immunogenicity and safety of the third dose booster immunization of Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01) in healthy participants immunized with two doses schedule of V-01.

The primary objective is to evaluate the Immunogenicity of the third dose booster immunization of V-01 in healthy participants immunized with two doses schedule of V-01.

The secondary objective is to evaluate the safety of the third dose booster immunization of V-01 in healthy participants immunized with two doses schedule of V-01.

DETAILED DESCRIPTION:
The plan is to booster immunize the participants previously in 10μg test group in V-01 clinical trial phase I, 48 participants are planned to be enrolled. The actual case number will be calculated by the participants who signed the ICF and got actual inoculation with the third dose.

Vaccination and follow-up:

Three to six months after the two doses of V-01 (10 μg) were vaccinated, the participants received a booster dose of investigational vaccine (V-01, 10 μg) at the deltoid muscle of the upper arm.

Perform safety and immunogenicity related inspections in accordance with the schedule in the plan.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the study and sign the informed consent form
* The participants who were enrolled in the 10 μg test group in the previous study titled "A Randomized, Double-blind, Placebo-controlled Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01) in Healthy Participants", and went through the full course immunization without meeting the exclusive criteria.
* No history of contact with confirmed, asymptomatic or suspected COVID-19 cases.
* Males of reproductive potential and females of childbearing potential voluntarily agree to take effective and acceptable contraceptive methods from the signing of informed consent form to 6 months after vaccination; females of childbearing age refer to premenopausal women and women within 2 years after menopause.

Exclusion Criteria:

* Innoculated with COVID-19 vaccines other than V-01;
* History of high fever (axillary temperature ≥ 39℃) and last for more than 3 days, or serious allergic reactions during the last immunization with V-01;
* History of obvious allergic reactions or allergic reactions that needed to be medical intervention during the last immunization with V-01;
* After two doses of V-01 inoculation, a newly diagnosed severe chronic disease or the original chronic disease is poorly controlled by drugs (applicable to ≥60 years old): history of chronic respiratory diseases (including moderate to severe asthma, COPD, pulmonary fibrosis) , Hypertension which can not be controlled by drugs (systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg), history of severe cardiovascular disease (including heart failure, coronary artery disease, cardiomyopathy), history of chronic kidney disease, history of cancer, diabetes (blood sugar) Unsatisfactory control or serious complications related to diabetes);
* Any confirmed or suspected immunosuppressive or immunodeficiency disorder, including HIV infection and asplenia; recurrent severe infections and administration of immunosuppressive drugs during the past 6 months, excluding topical steroids or short-term oral steroids (<14 days);
* Having received immunoglobulin and/or any blood products 3 months prior to the investigational vaccine dose;
* Other scenarios that may be medically, psychologically or socially contradicted with the trial protocol at the investigator's discretion or preclude informed consents of the participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-08-07 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Immunogenicity Endpoints | 14 days after booster immunization
  1. The seroconvension, GMT, and GMI of SARS-CoV-2 neutralizing antibodies (live virus, pseudovirus neutralizing test method)
  2. The seroconvension, GMT, and GMI of SARS-CoV-2 RBD antibodies (Enzyme-linked Immuno Sorbent Assay，ELISA)

SECONDARY OUTCOMES:
Safety Endpoints | Day 0-7 after booster immunization, 6 months after booster immunization
  1. The occurrence of AEs at each time point (at least 30 minutes, 0-7 days, and within 30 days after booster vaccination);
  2. The incidence of serious adverse events (SAE) (within 6 months after booster vaccination).

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Jikai, Principal Investigator — Guangdong Center for Disease Prevention and Control
Locations (1):
- Guangdong Provincial Center for Disease Control and Prevention, Guangzhou, Guangdong, China